CLINICAL TRIAL: NCT01788943
Title: Nicotinic Receptor Availability and Smoking Cessation Success.
Brief Title: Nicotine Receptor Levels and Smoking Cessation
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jacob Dubroff, Assistant Professor of Radiology, University of Pennsylvania
Other Study IDs: nAChR-PET-quit
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2017-08

CONDITIONS: Smoking Cessation; Nicotine Addiction
Keywords: positron emission tomography; nicotine receptor
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Slow metabolizers: Individuals with an NMR <0.26 will be classified as slow metabolizers.
- Normal metabolizers: Participants with an NMR >= 0.26 will be classified as normal metabolizers.

SUMMARY:
The investigators propose to use positron emission tomography (PET) imaging to determine whether nicotinic receptor availability at pretreatment predicts smoking cessation success. The investigators will recruit 30 smokers from those enrolled in the Pharmacogenetics of Nicotine Addiction Treatment clinical trial. The investigators will measure nicotinic receptor availability using the PET radioligand 2-[18F]FA, after overnight abstinence and prior to initiation of treatment.

DETAILED DESCRIPTION:
Subjects will be asked to complete a short screening session, an orientation phone call, and two imaging sessions: one PET imaging session and one MRI session.

Intake Session. This session will familiarize subjects with the study procedures and risks, as well as determine initial eligibility for the study. Subjects will first complete an Imaging Screening Form with study personnel. Subjects will also complete a Magnet Safety Form to check for any metal in the body. Finally, subjects will complete a Scanning Registration Form.

Orientation Call. Dr. Dubroff (the Principal Investigator and study physician) will call subjects before the PET Scan Session to review the study procedures and risks and answer any questions subjects might have.

PET Scan Session. Subjects will receive a telephone call the day before the session to remind them to stop smoking at 9:00pm that night. At the session, they will provide a series of samples. These include:

* A urine sample to assess for the presence of study-prohibited drugs and medications (including cocaine, opiates, benzodiazepines, amphetamines, methamphetamines, tri-cyclic antidepressants, methadone, PCP, and barbiturates).
* Women of childbearing age will be required to take a urine pregnancy test.
* A breath alcohol concentration (BrAC) measurement.
* A breath carbon monoxide (CO) reading.
* Have your weight measured.

After subjects arrive at the PET center, they will have two intravenous (I.V.) lines placed. A sterile solution will be dripped through the tubing to keep them open. Subjects will have blood pressure and heart rate taken prior to injection and three 10ml tubes of blood will be drawn to determine the baseline levels of radioactive tracer. After this, subjects will be injected with a radioactive tracer (a chemical that has a radioactive molecule attached to it) called 2-[18F]FA that will be pumped through one of the I.V. lines over an 8-hour period. During the waiting period subjects will complete two questionnaires, a brief IQ test, and five computer games. They will have repeated blood pressure and heart rate readings taken soon after the initial injection and every 45 minutes afterwards. The investigators will draw 3 ml (half a teaspoon) of blood from the second I.V. line every 15-30 minutes to measure radiotracer levels.

Just prior to beginning the scan, subjects will be asked two questions about cravings. These questions will be asked every 30 minutes during the scan and then once more after subjects have exited the scan. The investigators will draw one 3ml tube of blood at the beginning of the PET scan and every 30 min during the PET scan (total 5 teaspoons) from the second I.V. line to measure radiotracer levels.

ELIGIBILITY:
Exclusion Criteria:

In addition to the exclusion criteria used for PNAT trial [NCT01314001], participants in this trial will be excluded if they meet the following criteria:

Imaging-Related Exclusion Criteria:

1. Weigh over 299 lbs.
2. Self-reported history of head trauma or brain (or CNS) tumor.
3. Self-reported history of claustrophobia (contraindicated for PET and MRI).
4. Cochlear implant or bilateral hearing aids.
5. Pacemakers, certain metallic implants, or presence of metal in the eye as contraindicated for MRI.
6. History of gunshot wound (including BB guns).
7. Circumstances or conditions that may interfere with magnetic resonance imaging (MRI).
8. CO reading greater than 15ppm at the PET Scan Session (or at least a 50% reduction from the PNAT Intake Session).
9. BrAC reading greater than or equal to 0.01 at the PET Scan Session.
10. Positive urine drug screen for cocaine, phencyclidine, amphetamines, methamphetamines, tricyclic antidepressants, opiates, methadone, benzodiazepines, or barbiturates at the PNAT Intake Session or PET Scan Session.
11. Positive urine pregnancy (females only) screen at the PET Scan Session and/or MRI Scan Session.
12. Inability to give blood at the PET Scan Session (blood samples are required to analyze PET data).
13. Prior exposure to radioactive tracers in imaging studies or for medical reasons may be exclusionary.

General Exclusion Criteria:

1. Any medical condition, illness, disorder or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator or Co-investigators.
2. Inability to provide informed consent or complete the study procedures within 10 hours and/or correctly, as determined by the Principal Investigator or Co-investigators.
3. Any physical or visual impairment that would prevent completion of the cognitive tasks.
4. Participation (within the last 6 months) in other studies at our center involving similar cognitive testing procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  Participants will be male and female smokers between the ages of 18 and 65 and must be enrolled(consented and meet all eligibility requirements) in the ongoing PNAT trial [NCT01314001] in order to participate in this sub-study. They must be able to provide informed consent and weigh less than 300 lbs (due to limitations of the PET and MRI scanners).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brody AL, Mandelkern MA, London ED, Olmstead RE, Farahi J, Scheibal D, Jou J, Allen V, Tiongson E, Chefer SI, Koren AO, Mukhin AG. Cigarette smoking saturates brain alpha 4 beta 2 nicotinic acetylcholine receptors. Arch Gen Psychiatry. 2006 Aug;63(8):907-15. doi: 10.1001/archpsyc.63.8.907. PMID 16894067
- See also: Principal Investigator — http://www.med.upenn.edu/apps/faculty/index.php/g334/p6489091
- See also: Center for Interdisplinary Research on Nicotine Addiction — http://www.med.upenn.edu/cirna/
- See also: Position Emission Tomography (PET) Center at the University of Pennsylvania — http://www.uphs.upenn.edu/radiology/research/labs/pet-positron-emission-tomography/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10/01/2012-03/28/2014 recruitment at the Center for Interdisciplinary Research on Nicotine Addiction at the University of Pennsylvania
Groups:
- Slow Metabolizers.: Participants with an NMR < 0.26 will be considered slow metabolizers.
- Normal Metabolizers: Participants with an NMR >= 0.26 will be considered normal metabolizers.
Period: Overall Study
Arm/Group | Slow Metabolizers. | Normal Metabolizers
Started | 13 (Recruitment for study began.) | 12
Completed | 12 (2FA-PET Brain Image Analysis Completion Date) | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Nicotine Metabolizers: Nicotine Metabolite Radio of > or = 0.26
- Slow Nicotine Metabolizers: Nicotine Metabolite Radio of < 0.26.
- Total: Total of all reporting groups
Arm/Group | Normal Nicotine Metabolizers | Slow Nicotine Metabolizers | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Full Range); unit: years] | 48.7 [35 to 64] | 45.5 [23 to 62] | 47.1 [23 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Acetylcholinergic Nicotine Receptor Availability as Determined by 2FA -PET Brain Imaging.
Description: Acetylcholinergic Nicotine Receptor availability in the thalamus is decreased in smokers with slower rates of nicotine metabolism.
Time Frame: following overnight nicotine abstinence
Measure: Mean (Standard Deviation); unit: Distribution Volume Ratio (Vt/fp)
Groups:
- Slow Metabolizers.: Subjects with an NMR < 0.26.
- Normal Metabolizers: Subjects with an NMR of > or = 0.26.
Arm/Group | Slow Metabolizers. | Normal Metabolizers
Number analyzed (Participants) | 12 | 12
Distribution Volume Ratio (Vt/fp) | 17.5 (2.4) | 26.8 (3.1)
Statistical Analysis 1: Comparison: Slow Metabolizers. vs Normal Metabolizers; Test type: Other; p = 0.037, ANOVA

2. Secondary Outcome: Change in Cigarette Craving as Measured by the Questionnaire on Smoking Urges.
Description: Measure is post-scan subtracted from pre-scan ratings. Rating is measured using the standardized, Questionnaire on Smoking Urges - Brief Version (QSU-Brief) is a standardized measure consisting of 10 statements, each rated on a Likert-like scale from 1 (Strongly Disagree) to 7 (Strongly Agree). Responses for each item are summed to produce an overall score with a range of 10-70.
Time Frame: Before and immediately following the PET scan.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Slow Metabolizers. | Normal Metabolizers
Number analyzed (Participants) | 12 | 12
units on a scale | -8.1 (10.1) | 1.8 (7.7)
Statistical Analysis 1: Comparison: Slow Metabolizers. vs Normal Metabolizers; Test type: Other; p = 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events will examine the day of and the day following PET scanning.
Groups:
- Slow Metabolizers (NMR < 0.26); Normal Metabolizers (NMR > or + 0.26): No serious adverse events were observed.
Arm/Group | Slow Metabolizers (NMR < 0.26) | Normal Metabolizers (NMR > or + 0.26)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes